CLINICAL TRIAL: NCT01804010
Title: Pharmacokinetic, Pharmacodynamic Profiles and Safety After Oral Administration of Ivabradine in Male Healthy Korean Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Principal Investigator, Kyun-Seop Bae, Dep. of clinical pharmacology and therapeutics, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-0114
Record Dates: First submitted 2013-02-27; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Individual
MeSH Terms: interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivabradine (Active Comparator): Single and repeated oral administrations of 3 doses of ivabradine
  Interventions: Drug: Ivabradine and placebo
- Placebo (Placebo Comparator): Placebo administration
  Interventions: Drug: Ivabradine and placebo

INTERVENTIONS:
Drug: Ivabradine and placebo — Single and repeated oral administrations of 3 doses of ivabradine (2.5, 5, and 10 mg). Subjects were given a single administration of ivabradine during Period 1 (P1), following a 3-day washout, they were given repeated administrations twice daily for 4.5 days during Period 2 (P2).
  Other Names: Ivabradine; Placebo

SUMMARY:
1. To assess the pharmacokinetic profile of ivabradine (S 16257) and its main active metabolite S 18982 in Korean healthy volunteers after oral administration of ivabradine at the doses of 2.5, 5, 10mg and after repeated oral administrations of ivabradine for 4.5 days at the same doses twice daily versus placebo and to use the study results for bridging with Caucasian data.
2. The pharmacodynamic profile of ivabradine versus placebo by measuring its effects on heart rate after single and then after repeated administrations.
3. Clinical safety of ivabradine versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years and Korean
* Nonsmoker or smoke less than 5 cigarettes per day
* normal dietary habits
* BMI ranging from 18 to 25 kg/m2
* good physical and mental status, determined by the investigator
* vital signs in resting condition within range: SBP 100-139 mmHg, DBP 50-89 mmHg
* Normal ECG

Exclusion Criteria:

* Participate any other trial in the last 3 months prior to the study
* History of major psychiatric, medical, surgical disorders
* Acute, or chronic disease
* History of hypersensitivity to at least one drug
* History of alcoholism or positive alcohol breath test
* Positive drug screening results
* known positive serology for HIV1, HIV2, hepatitis B or C
* blood donor within the last 3 month of the study
* regular use of sedatives, hypnotics, tranquillisers

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Cmax,tmax, AUC(Area under the time-concentration curve) of ivabradine and metabolite | within 60 days after blood sampling (blood sample analysis)
  For PK measurements, blood samplings were done: pre-dose then 20 min, 40 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 36 h, 48 h, 60 h, and 72 h following the D1 single administration (P1) and the Day 8 (D8) last repeated dose (P2), respectively.Ivabradine and its main metabolite were determined using LC-MS/MS, then pharmacokinetic parameters were calculated by noncompartmental approach. Descriptive statistics were performed on the PK individual parameters calculated from the plasma concentration-time profiles.

SECONDARY OUTCOMES:
pharmacodynamics: The change of heart rate between baseline and over 24-hour, diurnal, nocturnal, awake, and asleep periods after administration of ivabradine | within 10 days after administration
  For PD measurements, 24-hour Holter recordings were performed on Day0, Day1, Day8, and Day10. a resting 12-lead ECG were also performed.
  The changes of heart rate between day 1 and baseline values, between day 8 and baseline values were studied over 24-hour, diurnal, nocturnal, awake and asleep period for each ivabradine dose in comparison with placebo. Descriptive statistics by dose were performed and confidence intervals of the differences between each dose of ivabradine and placebo were constructed using a non-parametric method based on Hodges & Lehman estimate for independent samples.

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea